CLINICAL TRIAL: NCT06188078
Title: The Effect of Bladder Stimulation Technique and Bathing Method on Urine Collection in Term Babies: A Randomized Controlled Trial
Brief Title: The Effect of Bladder Stimulation Technique and Bathing Method on Urine Collection in Term Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Zeynep Erkut, Assistant Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023/01-04
Record Dates: First submitted 2023-12-13; First posted 2024-01-03 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Urine Specimen Collection
Keywords: term babies; urine; bladder stimulation technique; bath
MeSH Terms: interventions — Baths

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): Babies in the control group will be fed only breast milk or formula, and a urine bag will be inserted after 25 minutes and they will be expected to urinate. The success of the transaction and the processing time will be recorded.
  Interventions: Other: Control
- The bladder stimulation technique (Experimental): Newborns will be fed formula or pumped breast milk, depending on the baby's age and weight. A urine bag will be inserted 25 minutes after the feeding.
  The newborn will be held under the armpit by the nurse, male infants will be held with their legs hanging down, and female infants will be held in the hip flexion position.
  Newborns with spontaneous voiding during the period from the beginning of the investigation procedure to positioning the newborn will be excluded from the study.
  The bladder stimulation technique will be repeated sequentially for 3 minutes until voiding begins.The success of the transaction and the processing time will be recorded.
  Interventions: Other: The bladder stimulation technique
- Bath (Experimental): Newborns will be fed formula or pumped breast milk, depending on the baby's age and weight. Babies will be bathed under running water 20 minutes after feeding.The bathing process will take 4 minutes in total. After bath, a urine bag will be inserted at the 25th minute of feeding. The success of the transaction and the processing time will be recorded.
  Interventions: Other: Bath

INTERVENTIONS:
Other: Control — Babies in the control group will be fed only breast milk or formula, and a urine bag will be inserted after 25 minutes and they will be expected to urinate. The success of the transaction and the processing time will be recorded.
  Arms: Control
Other: The bladder stimulation technique — Newborns will be fed formula or pumped breast milk, depending on the baby's age and weight. A urine bag will be inserted 25 minutes after the feeding.
  The newborn will be held under the armpit by the nurse, male infants will be held with their legs hanging down, and female infants will be held in the hip flexion position.
  Newborns with spontaneous voiding during the period from the beginning of the investigation procedure to positioning the newborn will be excluded from the study.
  The bladder stimulation technique will be repeated sequentially for 3 minutes until voiding begins.The success of the transaction and the processing time will be recorded.
  Arms: The bladder stimulation technique
Other: Bath — Newborns will be fed formula or pumped breast milk, depending on the baby's age and weight. Babies will be bathed under running water 20 minutes after feeding.The bathing process will take 4 minutes in total. After bath, a urine bag will be inserted at the 25th minute of feeding. The success of the transaction and the processing time will be recorded.
  Arms: Bath

SUMMARY:
Purpose of the Study: The aim of this study is to examine the effect of bladder stimulation technique and bathing method on urine collection in term infants hospitalized in the neonatal intensive care unit.

Content of the Study: This study will consist of 3 groups. Babies in the 1st group, the control group, will be fed only with breast milk or formula, and after 25 minutes, a urine bag will be inserted and urination will be expected. The babies in the second group, the bladder stimulation technique application group, will also be placed in a urine bag 25 minutes after feeding. Then the bladder stimulation technique will be applied. This technique; consists of two consecutive maneuvers. In the first maneuver, the bladder (Urine Bag) is stimulated by hitting the suprapubic (lower parts of the abdomen) area for 30 seconds at a frequency of 100 touches per minute. In the second maneuver, a 30-second circular massage is applied to the paravertebral region (located next to the spine). Babies in the 3rd group, the bathing group will be fed formula or pumped breast milk, depending on the baby's age and weight. Babies will be bathed under running water 20 minutes after feeding.The bathing process will take 4 minutes in total. After bath, a urine bag will be inserted at the 25th minute of feeding. In all group, urine urination will be monitored by running the stopwatch immediately after the urine bag is placed on all babies. When the baby urinates, the stopwatch will be stopped and the time and success of urination will be recorded on the observation form by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Term babies whose gestational age is 37+6 days and above,
* Full-term newborns aged 1-28 days
* Orally fed babies
* Babies with stable health status,
* Babies who do not have urological, neurological diseases, or anatomical anomalies that may affect bladder function,
* Babies of parents who voluntarily agree to participate in the study will be included in the study.

Exclusion Criteria:

* Preterm babies whose gestational age is below 37+6 days,
* Babies fed with an orogastric tube (OGS),
* Babies with serious health problems (such as respiratory distress),
* Babies with urological, neurological diseases or anatomical anomalies that may affect bladder function,
* Babies of parents who do not agree to participate in the study will be excluded from the study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Success in Urination | During the procedure (3 minutes)
  Success in urination is defined as urine sample collection within 3 minutes (180 seconds)
Total Urination Time | During the procedure (3 minutes)
  Total urination time is defined as the time elapsed from the urine collection collector bag placed on the baby to the beginning of the micturition.

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University, Istanbul, Turkey (Türkiye)